CLINICAL TRIAL: NCT00117104
Title: A Multicenter Study Evaluating Once Weekly Intravenous Administration of Aranesp® in Subjects With End Stage Renal Disease on Chronic Hemodialysis
Brief Title: Evaluating Aranesp® in Subjects With End Stage Renal Disease onChronic Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030133
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease (ESRD); Kidney Disease, Dialysis; Aranesp®, rHuEPO; Anemia, Hemoglobin; Dosing, Amgen
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
The purpose of this study is to assess the Aranesp® dose administered intravenously (IV) once weekly to maintain hemoglobin (Hgb) levels in hemodialysis subjects who are either recombinant human erythropoietin (rHuEPO) naïve or subjects converted from rHuEPO therapy administered IV thrice weekly (TIW).

ELIGIBILITY:
Inclusion Criteria: - Subjects with end stage renal disease (ESRD) on hemodialysis Exclusion Criteria: - Known hypersensitivity to Aranesp® (darbepoetin alfa) or any of its excipients - Participating in an investigational drug or device trial - Patient will not be available for follow-up assessment - Patient has any disorder that compromises the ability of the patient to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Target hemoglobin (Hgb)

SECONDARY OUTCOMES:
Distribution of hemoglobin (Hgb) values by week

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com